CLINICAL TRIAL: NCT00764946
Title: A Phase III Open-Label Single Arm Study to Evaluate the Safety, Tolerability, and Efficacy of MK0518/Raltegravir in a Diverse Cohort of HIV-Infected Patients
Brief Title: A Study of Raltegravir in a Diverse Cohort of HIV-Infected Patients (0518-055)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0518-055; 2008_555
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

ARMS (1):
- 1 (Experimental): raltegravir
  Interventions: Drug: Comparator: raltegravir

INTERVENTIONS:
Drug: Comparator: raltegravir — 400 mg tablets taken twice daily. Total treatment period is 48 weeks.
  Other Names: ISENTRESS

SUMMARY:
A study to test the safety and effect of twice daily raltegravir in a diverse cohort of patients currently infected with human immunodeficiency virus (HIV), where at least 50% are African American and at least 25% are female, either having received antiretroviral drugs before or not.

ELIGIBILITY:
Inclusion Criteria:

* Patient is HIV positive
* Patient agrees to use (or have their partner use) birth control as defined by the study doctor

Exclusion Criteria:

* If female, pregnant or breastfeeding
* Patient has used an investigational agent in the last 30 days
* Patient has acute hepatitis
* Patient has received MK0518 (raltegravir) before
* Patient has used another experimental HIV-integrase inhibitor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Squires KE, Bekker LG, Eron JJ, Cheng B, Rockstroh JK, Marquez F, Kumar P, Thompson M, Campo RE, Mounzer K, Strohmaier KM, Lu C, Rodgers A, Jackson BE, Wenning LA, Robertson M, Nguyen BY, Sklar P; REALMRK Investigators. Safety, tolerability, and efficacy of raltegravir in a diverse cohort of HIV-infected patients: 48-week results from the REALMRK Study. AIDS Res Hum Retroviruses. 2013 Jun;29(6):859-70. doi: 10.1089/AID.2012.0292. Epub 2013 Feb 26. PMID 23351187

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Failing Current Therapy: Participants with previous HIV treatment experience who did not respond to their current HIV therapy were treated with open-label raltegravir 400 mg twice daily (b.i.d.) plus other antiretroviral agents at the discretion of the investigator.
- Participants Intolerant to Current Therapy: Participants with previous HIV treatment experience who could not tolerate the treatment were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
- Participants Treatment Naive: Participants with no previous HIV treatment were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
Period: Overall Study
Arm/Group | Participants Failing Current Therapy | Participants Intolerant to Current Therapy | Participants Treatment Naive
Started | 98 | 89 | 22
TREATED | 97 | 88 | 21
Completed | 85 | 72 | 18
Not Completed | 13 | 17 | 4
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0
Not completed — Physician Decision | 2 | 4 | 0
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 6 | 2
Not completed — Never Treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Failing Current Therapy: Participants with previous HIV treatment experience who did not respond to their current HIV therapy were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
- Total: Total of all reporting groups
Arm/Group | Participants Failing Current Therapy | Participants Intolerant to Current Therapy | Participants Treatment Naive | Total
Number analyzed (Participants) | 97 | 88 | 21 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants who did not receive treatment are excluded from this measure.
  years | 44.0 (9.2) | 46.9 (9.0) | 38.5 (10.1) | 44.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants who did not receive treatment are excluded from this measure.
  Participants
    Female | 46 | 44 | 7 | 97
    Male | 51 | 44 | 14 | 109
Race [Number; unit: Participants] — Participants who did not receive treatment are excluded from this measure.
  Participants
    Black | 70 | 69 | 14 | 153
    Non-Black | 27 | 19 | 7 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved HIV Ribonucleic Acid (RNA) <50 Copies/mL at Week 48
Description: Numbers of participants with HIV RNA copies <50 copies/mL were summarized by race for each time point.
Time Frame: Week 48
Population: Efficacy analyses were based on the Full Analysis Set population that included all participants who took at least one dose of study medication and had at least one postbaseline evaluation.
  The Treatment-Related Discontinuation = Failure approach was used as the primary method for handling missing HIV RNA values.
Measure: Number; unit: Participants
Groups:
- Treatment Experienced - Failing Current Therapy: Participants with previous HIV treatment who did not respond to their current HIV therapy were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
- Treatment Experienced - Treatment Intolerant: Participants with previous HIV treatment experience who could not tolerate their current HIV therapy were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
- Treatment Naive: Participants with no previous HIV treatment experience were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Treatment Intolerant | Treatment Naive
Number analyzed (Participants) | 94 | 80 | 21
Participants
  Black (n = 69, 62, 14) | 44 | 43 | 11
  Non-Black (n = 25, 18, 7) | 16 | 18 | 5

2. Secondary Outcome: Number of Participants Who Achieved HIV RNA <400 Copies/mL at Week 48
Description: Numbers of participants with HIV RNA copies <400 copies/mL were summarized by race for each time point.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment-Experienced - Treatment Intolerant | Treatment Naive
Number analyzed (Participants) | 94 | 81 | 21
Participants
  Black (n = 69, 62, 14) | 51 | 50 | 12
  Non-Black (n = 25, 18, 7) | 17 | 18 | 5

3. Secondary Outcome: Mean Change From Baseline to Week 48 in HIV RNA
Description: Mean changes from baseline in plasma HIV RNA were summarized by race at each time point.
Time Frame: Baseline and Week 48
Population: Efficacy analyses were based on the Full Analysis Set population that included all participants who took at least one dose of study medication and had baseline and at least one postbaseline evaluation.
  Baseline values were carried forward for participants who discontinued before Week 48 due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Groups:
- Treatment Experienced - Failing Current Therapy: Participants with previous HIV treatment experience who did not respond to their current HIV therapy were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
- Treatment Naive: Participants with no previous HIV treatment were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Treatment Intolerant | Treatment Naive
Number analyzed (Participants) | 77 | 22 | 19
log10 copies/mL
  Black (n = 55, 16, 13) | -1.62 [-1.93 to -1.31] | -1.16 [-1.88 to -0.45] | -2.49 [-3.17 to -1.81]
  Non-Black ( n= 22, 6, 6) | -1.52 [-2.05 to -0.99] | -2.21 [-2.87 to -1.56] | -1.66 [-3.14 to -0.18]

4. Secondary Outcome: Mean Change From Baseline to Week 48 in CD4 Cell Count
Description: Mean changes from baseline in CD4 cell counts were summarized by race at each time point.
Time Frame: Baseline and Week 48
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Treatment Intolerant | Treatment Naive
Number analyzed (Participants) | 89 | 76 | 19
cells/mm^3
  Black (n = 66, 61, 12) | 141.0 [109.6 to 172.5] | 62.3 [27.0 to 97.7] | 208.8 [108.6 to 309.1]
  Non-Black (n = 23, 15, 7) | 113.1 [62.2 to 164.1] | 69.2 [16.7 to 121.7] | 164.4 [12.8 to 316.1]

5. Secondary Outcome: Number of Participants Without Loss of Virologic Response
Description: For participants with confirmed HIV RNA levels <50 copies/mL on 2 consecutive visits, loss of virologic response is the occurrence of the first value >50 copies/mL or loss to follow-up; participants who never achieved HIV RNA <50 copies/mL on 2 consecutive visits are also considered as having loss of virologic response. Events are the numbers of participants with loss of virologic response versus the numbers of participants with no loss of virologic response (event free).
Time Frame: Week 48
Population: Efficacy analyses were based on the Full Analysis Set population that included all participants who took at least one dose of study medication and had at least one postbaseline evaluation.
Measure: Number; unit: participants
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Treatment Intolerant | Treatment Naive
Number analyzed (Participants) | 97 | 88 | 21
participants
  Black (n = 70, 69, 14) | 48 | 49 | 11
  Non-Black (n = 27, 19, 7) | 16 | 17 | 5

6. Primary Outcome: Number of Participants With One or More Adverse Events
Description: Numbers of participants with one or more adverse events were summarized by race.
Time Frame: Week 48
Measure: Number; unit: Participants
Groups:
- Treatment Experienced - Intolerant To Current Therapy: Participants with previous HIV treatment experience who could not tolerate their current HIV therapy were treated with open-label raltegravir 400 mg b.i.d. plus other antiretroviral agents at the discretion of the investigator.
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Intolerant To Current Therapy | Treatment Naive
Number analyzed (Participants) | 97 | 88 | 21
Participants
  Black (n = 70, 69, 14) | 55 | 40 | 12
  Non-Black (n = 27, 19, 7) | 23 | 13 | 6

7. Primary Outcome: Number of Participants Who Discontinued Due to an Adverse Event
Description: Numbers of participants who discontinued due to an adverse event were summarized by race.
Time Frame: Week 48
Measure: Number; unit: Participants
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Intolerant To Current Therapy | Treatment Naive
Number analyzed (Participants) | 97 | 88 | 21
Participants
  Black (n = 70, 69, 14) | 1 | 2 | 1
  Non-black (n = 27, 19, 7) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment Experienced - Failing Current Therapy | Treatment Experienced - Intolerant To Current Therapy | Treatment Naive
Serious Adverse Events (participants affected / at risk) | 15/97 | 5/88 | 2/21
Other Adverse Events (participants affected / at risk) | 49/97 | 26/88 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Experienced - Failing Current Therapy (N=97) | Treatment Experienced - Intolerant To Current Therapy (N=88) | Treatment Naive (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sensorineural hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Acute gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Community acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Depression worsened (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Experienced - Failing Current Therapy (N=97) | Treatment Experienced - Intolerant To Current Therapy (N=88) | Treatment Naive (N=21)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (18) | 7 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (13) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 5 (6) | 2 (2) | 0 (0)
Common cold (Infections and infestations) | 5 (6) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 8 (10) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 9 (10) | 2 (2)
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Twenty-four months after completion of this study or after publication of the multicenter results, an investigator may publish the results for their study site independently. The sponsor must have the opportunity to review all proposed publications or presentations regarding the study 60 days before submission.